CLINICAL TRIAL: NCT06043388
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial to Evaluate the Safety and Tolerability of Omicron BA.4/5-Delta Strain Recombinant Novel Coronavirus Protein Vaccine (CHO Cells) in People Aged 18 Years and Above.
Brief Title: Omicron BA.4/5-Delta COVID-19 Vaccine Phase I Clinical Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Hunan Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2023-NCV-V04
Record Dates: First submitted 2023-08-31; First posted 2023-09-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cell)
  Interventions: Biological: Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells)
- Group 2 (Placebo Comparator): physiological saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) — Inoculate one dose, 0.5ml，Intramuscular injection into the deltoid muscle of the upper arm
  Arms: Group 1
Biological: Placebo — Inoculate one dose, 0.5ml，Intramuscular injection into the deltoid muscle of the upper arm
  Arms: Group 2

SUMMARY:
The purpose of this study is to evaluate the safety of Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) after vaccination in people aged 18 and over. It is planned to screen 100 subjects who are 18 years old and above and more than 6 months since the last new coronavirus infection or new coronavirus vaccine. All subjects collected venous blood before vaccination, 14 days, 3 months, and 6 months after vaccination for immunological detection of neutralizing antibody of the new coronavirus prototype strain, Delta strain and Omicron strain (BA.4/5, XBB); All adverse events (AEs) within 30 minutes after vaccination, all AEs (including solicited and non-solicited AEs) on days 0-7, all AEs (non-solicited AEs) on days 8-30, and all AEs within 12 months after vaccination were collected. serious adverse events (SAE) and adverse events of special interest (AESI).

DETAILED DESCRIPTION:
Solicitation AEs (the following events occurring within 7 days of vaccination):

AESI:

Select 100 cases of people aged 18 years and above and more than 6 months after the last new coronavirus infection or vaccination, and evaluate the effectiveness of Omicron BA.4/5-Delta strain recombinant new coronavirus protein vaccine (CHO cells) in people aged 18 years and above. Safety after vaccination in the population.

Non-vaccination site (systemic) adverse events: fever, headache, fatigue/asthenia, nausea, vomiting, diarrhea, myalgia (non-vaccination site), cough, acute allergic reaction.

Venous blood was collected from all subjects before vaccination, 14 days, 3 months, and 6 months after vaccination for immunological detection of neutralizing antibodies against the new coronavirus prototype strain, Delta strain, and Omicron strain (BA.4/5, XBB).

Adverse events at the vaccination site (local): pain, swelling, induration, redness, rash, itching; Myocarditis/pericarditis, thrombosis, thrombocytopenia, etc., immune-related diseases (psoriasis, rheumatoid arthritis, etc.), nervous system-related diseases (Glibari syndrome, peripheral neuropathy, Bell's palsy).

Pregnancy events that occurred within 12 months after vaccination of subjects in this trial were collected, and neonates whose pregnancy outcome was delivery during the study period were followed up for long-term safety (follow-up until 12 months after delivery).

Immunogenicity observation:

Safety observations:

AEs, AESIs and SAEs: collect all adverse events (AEs) 30 minutes after vaccination, all AEs 0-7 days (including solicited and non-solicited AEs), 8-30 days all AEs (non-solicited AEs), vaccination All serious adverse events (SAEs) and adverse events of special interest (AESIs) within the last 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above when signing the informed consent form;
* The subject himself voluntarily participates in this research, and signs the informed consent form, and can provide legal identification, understand and abide by the requirements of the trial protocol;
* Female subjects of childbearing age and male subjects must agree to take effective contraceptive measures during the study.

Exclusion Criteria:

* Less than 6 months since the last COVID-19 infection or COVID-19 vaccination；
* Prior history of severe allergy to any vaccine, or to any component of the experimental vaccine, including aluminum preparations, such as anaphylactic shock, allergic laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, dyspnea, angioneurotic edema, allergy (such as allergy to two or more drugs, food or pollen);
* Suspected or confirmed fever (axillary temperature ≥37.3℃/ mouth temperature ≥37.5℃) within 72 hours before enrollment, or axillary body temperature ≥37.3℃/ mouth temperature ≥37.5℃ on the day of enrollment;
* Patients with uncontrolled lymphoproliferative disease, unmitigated aplastic anemia, primary immune thrombocytopenia (ITP) activity, uncontrolled coagulation disease, etc.;
* a history of congenital or acquired immunodeficiency or autoimmune disease; Absence of spleen, or history of splenic surgery, trauma or immunomodulator treatment within 6 months, such as immunosuppressive dose of glucocorticoids (dose reference: equivalent to prednisone 20mg/ day for more than a week); Or monoclonal antibodies; Thymosin; Or interferon; Topical use (such as ointments, eye drops, inhalants or nasal sprays) is permitted;
* Non-live vaccine should be administered within 14 days before vaccination, and live attenuated vaccine should be administered within 30 days;
* Patients with malignant tumors who are undergoing chemotherapy, radiotherapy, immunotherapy, etc., before and after surgery; Patients with organ transplant status;
* People with uncontrolled epilepsy and other progressive neurological disorders (e.g. Transverse myelitis, Guillain-Barre syndrome, demyelinating diseases, etc.);
* Patients with acute disease, or acute onset of chronic disease, or uncontrolled severe chronic disease, such as medically uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg);
* Participants who had used blood and blood-related products within 3 months prior to enrollment;
* Participants who have participated in or are participating in other clinical trials (including drugs and devices) within 3 months prior to the clinical trial;
* Women of childbearing age have had unprotected sexual activity within 14 days prior to enrollment
* lactating women or women during pregnancy;
* The investigator determined that the subject had any disease or condition that would put the subject at risk, that the subject would not be able to complete the trial as required by the protocol, or that there would be conditions that would interfere with the evaluation of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint | Within 12 months after vaccination
  Incidence of AEs&SAE&AESI

SECONDARY OUTCOMES:
Immunogenicity endpoint | 14 days after vaccination
  Geometric mean titer (GMT) of SARS-CoV-2 neutralizing antibody

CONTACTS AND LOCATIONS:
Overall Officials: Junshi Zhao, Master, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention

IPD SHARING:
Plan to Share IPD: No